CLINICAL TRIAL: NCT04982926
Title: A Phase 1 Study of TAS2940 in Patients With Locally Advanced or Metastatic Solid Tumors With EGFR and / or HER2 Aberrations
Brief Title: A Study of TAS2940 in Participants With Locally Advanced or Metastatic Solid Tumor Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After careful review of Taiho's ongoing portfolio and data obtained so far in the context of broader landscape of clinical development in NSCLC HER2mut, Sponsor has made a strategic decision to terminate this study and not based on safety concerns.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAS2940-101; 2021-002189-41 (EudraCT Number)
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor; Glioblastoma; Non-small Cell Lung Cancer; Breast Cancer
MeSH Terms: conditions — Glioblastoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TAS2940 Dose Escalation (Experimental): Dose escalation will assess the safety and determine the maximum tolerated dose, the recommended phase 2 dose and the recommended dosing regimen of TAS2940 administered orally.
  Interventions: Drug: TAS2940
- Dose Expansion Non-small Cell Lung Cancer (Experimental): Dose expansion will assess preliminary anti-tumor activity in select solid tumors characterized by HER2 or EGFR aberrations
  Interventions: Drug: TAS2940
- Dose Expansion Breast Cancer (Experimental): Dose expansion will assess preliminary anti-tumor activity in select solid tumors characterized by HER2 or EGFR aberrations
  Interventions: Drug: TAS2940
- Dose Expansion Gliblastoma (Experimental): Dose expansion will assess preliminary anti-tumor activity in select solid tumors characterized by HER2 or EGFR aberrations.
  Interventions: Drug: TAS2940
- Dose Expansion Solid tumors (Experimental): Dose expansion will assess preliminary anti-tumor activity in select solid tumors characterized by HER2 or EGFR aberrations.
  Interventions: Drug: TAS2940

INTERVENTIONS:
Drug: TAS2940 — Study participants with solid tumors and EGFR or HER2 aberrations will receive TAS2940 tablets daily at increasing doses until MTD is reached.
  Arms: TAS2940 Dose Escalation
Drug: TAS2940 — Study subjects with select solid tumors characterized by EGFR or HER2 aberrations will receive TAS2940 at the dose identified during Dose Escalation phase.
  Arms: Dose Expansion Breast Cancer; Dose Expansion Gliblastoma; Dose Expansion Non-small Cell Lung Cancer; Dose Expansion Solid tumors

SUMMARY:
This is a first-in-human, open label, multicenter study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and the preliminary antitumor activity of TAS2940 in patients with advanced or metastatic solid tumors who are not candidates for approved or available therapies.

DETAILED DESCRIPTION:
TAS2940 is a small molecule inhibitor of ERBB family proteins HER2 and EGFR. It has not been evaluated in human subjects yet. The study will be conducted in 2 parts, dose escalation and dose expansion. The dose escalation part will assess the safety and determine the maximum tolerated dose, the recommended phase 2 dose and the recommended dosing regimen of TAS2940 administered orally. The dose expansion part will assess preliminary anti-tumor activity in select solid tumors characterized by HER2 or EGFR aberrations.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed solid cancer that is locally advanced and metastatic and available standard treatment options have been exhausted
* Have adequate organ function
* ECOG PS 0-1

Dose Escalation:

* Have measurable or non- measurable disease per RECIST criteria v1.1 or RANO
* Any solid tumor with EGFR and / or HER2 aberration

Dose Expansion:

* Have measurable disease per RECIST criteria v1.1 for solid tumor (excluding primary brain tumor) or RANO (for glioblastoma)
* Cohort A: Non-small cell lung cancer (NSCLC)
* Cohort B: HER2 positive breast cancer
* Cohort C: Recurrent or refractory glioblastoma
* Cohort D: Other solid tumors with EGFR or HER2 aberrations

Exclusion Criteria:

* Non-stable brain metastases
* Have significant cardiovascular disorder
* Have not recovered from prior cancer treatment
* A serious illness or medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Dose Escalation:Maximum Tolerated Dose (MTD) | One Month
  Determine the incidence of dose-liming toxicities (DLTs) and adverse events (AEs) graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 within the first cycle
Dose Expansion:Overall Response Rate | 6 Months
  Document the ORR, defined as proportion of patients experiencing a best overall response of Complete Response (CR) or Partial response (PR) based on investigator accessed radiographic response per RECIST 1.1 or RANO criteria

SECONDARY OUTCOMES:
Dose Escalation: Overall Response Rate (ORR) | 6 Months
  Document the ORR defined as proportion of patients experiencing a best overall response of Complete Response (CR) or Partial response (PR) based on investigator accessed radiographic response per RECIST 1.1 or RANO criteria
Dose Escalation:Pharmacokinetic (PK) Profile | 3 Months
  Evaluation of the maximum observed plasma concentration; time to reach maximum concentration, area under the Concentration-time curve and time it takes for plasma concentration to fall by half its original value (T1/2) of TAS2940
Dose Expansion:Incidence of treatment-emergent Adverse Events (Safety and tolerability) | Estimated up to 6 months
  Safety and tolerability of TAS2940 based on reported AEs, graded according to NCI-CTCAE v.5.0
Dose Expansion:Duration of Response (DOR) | Estimated up to 6 months
  DOR, defined as time from the first documentation of response to date of objective tumor progression or death due to any cause, whichever occurs first.
Dose Expansion:Disease Control Rate (DCR) | Estimated up to 6 months
  DCR, defined as the proportion of patients experiencing a best overall response of Stable Disease (SD), PR or CR
Dose Expansion:Progression Free Survival (PFS) | Estimated up to 6 months
  Date of PR or CR to date of objective progression or death due to any cause.
Dose Expansion:Pharmacokinetic profile of TAS2940 | 3 Months
  Evaluation of the maximum observed plasma concentration; time to reach maximum concentration, area under the Concentration-time curve and time it takes for plasma concentration to fall by half its original value (T1/2) of TAS2940

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- CLCC Gustave Roussy, Villejuif, Cedex, France

IPD SHARING:
Plan to Share IPD: No